CLINICAL TRIAL: NCT02307942
Title: Does Intense Weight Loss Improve Physical Performance in Obese Patients Older Than 60 Yrs Undergoing Exercise Training? Comparison Between Surgery and Standard of Care.
Brief Title: Improvement in Physical Performance and Obesity Surgery in Patients Older Than 60 Years
Acronym: ELDSURG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13 7051 01; 13705101 (Other Grant/Funding Number: PHRC National 2013)
Record Dates: First submitted 2014-09-16; First posted 2014-12-04 (Estimated); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Obesity
Keywords: Randomized Clinical Trials; gastric banding; calorie restriction; SPPB; physical performance; elderly
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SURGERY (Experimental): Patient will be operated for a gastric banding disposal
  Interventions: Procedure: Gastric banding
- STANDARD (No Intervention): Standard of care for obesity

INTERVENTIONS:
Procedure: Gastric banding — The bariatric procedure is a gastric banding under general anesthesia with all the centres using the same surgical procedure (harmonized by group meetings). The laparoscopic surgical procedure has been described. The ERAS protocol will be applied in each centre. The inflation of the band will follow the procedures described by 0'Brien. The patients will attend a group education session before surgery, during which the eating behaviour with a band will be explained and practiced. Then after surgery, the routine procedure is applied.
  Arms: SURGERY

SUMMARY:
The main objective of this study is to compare the efficacy of two weight losing strategies (obesity surgery with gastric banding, and standard of care) on physical performance in elderly obese persons submitted to a physical training. Our hypothesis is that a surgery-induced weight loss in the context of a physical training (which is recommended in people 60-75 yrs losing weight) improves physical performance as compared to standard of care (3-5% weight loss).

DETAILED DESCRIPTION:
Randomized clinical trial; Single Blind A physical training is recommended in people above 60 yrs. engaged in a weight-losing program, in order to prevent the impairment of physical performance. Therefore a physical training program (endurance and strength training) will be implemented for all subjects participating in the study, starting 1 month before randomization. It will last for 13 months. Patients will be randomized either in the surgical group (gastric banding under general anesthesia) or in the reference group (mild calorie restriction and coaching). Physical performance of patients is evaluated at screening, inclusion, at randomization, 6 and 12 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

Criteria specific to the study Subjects aged 60 or over and younger than 75 yrs., seeking obesity treatments, seeking obesity surgery, with a BMI of 30 kg/m² or more, with comorbidities (see below), and a mildly decreased physical performance (SPPB between 5 and 8) are considered to participate in the study Criteria specific to obesity surgery This projects extends the classical recommendation for obesity surgery to people with a BMI of 30 and over with either the comorbidities list below, or a SPPB between 5 and 8. This level of physical impairment can be considered as a comorbidity in the elderly.

The French Ministry of health (HAS) recommends that obesity surgery be considered (here with a gastric banding) in patients fulfilling the following criteria:

* Subjects with a BMI of 40kg/m² or more, or 35kg/m² or more if at least one comorbidity that can be improved by weight loss is present among hypertension, obstructive sleep apnea, severe metabolic disorder (such as type 2 diabetes, NASH), or rheumatologic conditions associated with disability.
* After the failure of well designed medical, dietetic, psychological intervention followed up for 6-12 months, with no sufficient weight loss or in case of the failure of maintaining weight loss
* In subjects well informed of the consequences of surgery, and after a multi-disciplinary evaluation
* Subjects have understood and accepted the need for a long term medical and surgical follow up
* The risk of surgery is acceptable
* patient who signed the informed consent
* patient affiliated to a social security cover or equivalent

Exclusion Criteria:

Criteria specific to the study

* These are the impossibility to follow a physical training (unstable coronary heart disease, severe lung function impairment, rheumatologic conditions preventing training, a SPPB score below 5, cancer treatment within the 3 last months, Parkinson's disease, other severe illness that may interfere with physical activity) Criteria specific to gastric banding
* Cognitive impairment (MMSE ≤ 25)
* Severe eating disorder
* Impossible long-term follow-up
* Alcohol or drug dependence
* Lack of previous well designed obesity care
* Vital prognosis engaged in the short term
* Contra-indications to anaesthesia Classical criteria for the non inclusion in a trial
* The subject is in jail, or has freedom restriction
* Guardianship curators or judicial protection
* Patients participating in another intervention study.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-07-29 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-04 (Actual)

PRIMARY OUTCOMES:
Physical performance | 12 months, comparing to the 6 months assesment
  Short Physical Performance Battery score (SPPB)

SECONDARY OUTCOMES:
Physical performance | At randomization, 6 and 12 months later
  the components of the SPPB score
weight loss | At randomization, 6 and 12 months later
  kg, and % of initial weight
Composition of weight loss | At randomization, 6 and 12 months later
  % of weight lost as lean mass, as fat mass, changes in appendicular skeletal muscle mass
Changes in muscle strength | At randomization, 6 and 12 months later
  strain gauge
Changes in aerobic fitness | At randomization, 6 and 12 months later
  maximal aerobic capacity
Early complications | At randomization, 6 and 12 months later
  in operated patients : number of hospital re-admissions, number of deep venous thrombosis, number of pulmonary embolism, food intake (calories, protein, eating difficulties
Calorie and protein intake | At randomization, 6 and 12 months later
  dietary survey
Quality of life score | At randomization, 6 and 12 months later
  Nottingham quality of life score
Disability | At randomization, 6 and 12 months later
  Functional Status Questionnaire score
Cognitive function | At randomization, 6 and 12 months later
  MMSE

CONTACTS AND LOCATIONS:
Overall Officials: Patrick RITZ, MD; PhD, Principal Investigator — University Hospital of Toulouse, France
Locations (7):
- France (7):
  - Clinique de l'ANJOU, Angers
  - Hôpital louis Mourier, Colombes
  - CHU de LILLE, Lille
  - Hospices Civils de LYON, Lyon
  - CHU de Nantes, Nantes
  - HEGP, Paris
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Background] Chevallier JM, Zinzindohoue F, Douard R, Blanche JP, Berta JL, Altman JJ, Cugnenc PH. Complications after laparoscopic adjustable gastric banding for morbid obesity: experience with 1,000 patients over 7 years. Obes Surg. 2004 Mar;14(3):407-14. doi: 10.1381/096089204322917954. PMID 15072664
- [Background] O'Brien PE, MacDonald L, Anderson M, Brennan L, Brown WA. Long-term outcomes after bariatric surgery: fifteen-year follow-up of adjustable gastric banding and a systematic review of the bariatric surgical literature. Ann Surg. 2013 Jan;257(1):87-94. doi: 10.1097/SLA.0b013e31827b6c02. PMID 23235396
- [Background] Mittermair RP, Obermuller S, Perathoner A, Sieb M, Aigner F, Margreiter R. Results and complications after Swedish adjustable gastric banding-10 years experience. Obes Surg. 2009 Dec;19(12):1636-41. doi: 10.1007/s11695-009-9967-7. PMID 19763708
- [Background] Chevallier JM, Paita M, Rodde-Dunet MH, Marty M, Nogues F, Slim K, Basdevant A. Predictive factors of outcome after gastric banding: a nationwide survey on the role of center activity and patients' behavior. Ann Surg. 2007 Dec;246(6):1034-9. doi: 10.1097/SLA.0b013e31813e8a56. PMID 18043107
- [Background] Gagner M, Milone L, Yung E, Broseus A, Gumbs AA. Causes of early mortality after laparoscopic adjustable gastric banding. J Am Coll Surg. 2008 Apr;206(4):664-9. doi: 10.1016/j.jamcollsurg.2007.11.014. Epub 2008 Jan 28. PMID 18387472